CLINICAL TRIAL: NCT05046210
Title: Oral Exercise With Lay Health Advisor Strategy on Oral Self-care Behaviors, Oral Hygiene, Oral Function and Quality of Life Among Older Adults in Aboriginal Communities in Taiwan: A Randomized Controlled Trial
Brief Title: The Effectiveness of Lay Health Advisors Strategy Intervention on Aborigines Elderly Oral Care Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-SV(I)-20190010; NHRI-108A1-PHCO-03191908 (Other Grant/Funding Number: National Health Research Institutes (NHRI))
Record Dates: First submitted 2021-08-27; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Oral Health
Keywords: Aboriginal; Lay Health Advisor; Oral Hygiene; Quality of Life; Oral Function

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial (RCT) was conducted. The participants recruited from aboriginal communities in Eastern Taiwan. Data collecting time was from 2019 to 2020. Participants from the identified communities were randomly assigned to experimental group or control group using random table.
Who Masked: Participant
Masking Description: Participants from the identified communities were randomly assigned to experimental group or control group using random table.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LHA group (EG) (Experimental): Behavioral: LHA intervention
  Oral exercise intervention is designed to increase the range of movement in tongue, lips, and jaw as well as salivary gland massages, which will help speech and/or swallow functioning. All participants performed oral exercise before three meals a day, whereas the participants in the EG also received 4 lessons from a LHA over 4 weeks.
  Interventions: Behavioral: LHA intervention; Behavioral: Oral exercise intervention
- Leaflet group (CG) (Placebo Comparator): Oral exercise intervention is designed to increase the range of movement in tongue, lips, and jaw as well as salivary gland massages, which will help speech and/or swallow functioning. All participants performed oral exercise before three meals a day.
  The participants in the CG received oral exercise intervention and leaflets only.
  Interventions: Behavioral: Oral exercise intervention

INTERVENTIONS:
Behavioral: LHA intervention — The participants in the EG received 4 lessons from a LHA over 4 weeks. Four lessons were taught one-on-one once a week by a certified LHA at the participants' homes. The lessons including understand oral structure, learn oral self-care skills and oral function promotion, understand the status of oral self-care and the relationship between oral diseases and systemic diseases, understand swallowing dysfunction and safe eating skills and review.
  Arms: LHA group (EG)
Behavioral: Oral exercise intervention — Oral exercise intervention is designed to increase the range of movement in tongue, lips, and jaw as well as salivary gland massages, which will help speech and/or swallow functioning. All participants performed oral exercise before three meals a day.

SUMMARY:
In the present study, the investigators aimed to evaluate the effectiveness of community-based oral exercise with LHA intervention on the oral health-related quality of life, oral function and oral self-care behaviors. This randomized controlled trial included LHA group (EG) and leaflet group (CG), respectively. The EG received a four-week one-on-one session by an LHA. Baseline and follow-up data collection were used to collect the data in oral Self-care behaviors, oral hygiene, oral function and quality of life.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) was conducted. The participants recruited from aboriginal communities in Eastern Taiwan. Data collecting time was from 2019 to 2020. Participants from the identified communities were randomly assigned to EG or CG using random table. Participants who were 55 years old or above and indigenous people were recruited in the study. Participants who were disability, have had oral cancer, impaired facial appearance and impaired cognitive function were excluded. Impaired cognitive function was screening by Short Portable Mental Status Questionnaire (SPMSQ). Participants were recruited according to the predetermined minimal sample size estimated based on a type I error = 0.05, power = 0.95, and effect size (ES) f = 0.25 (medium effect in Cohen's f) . The number of samples in each group was expected 66 participants. An additional 30% drop out rate was added. The final number of samples for each group were required at least 86 participants. The total sample size was 122 and 118 in EG and CG, respectively. All participants underwent data collection at baseline and at 2-week, 3-and 6-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* 55 years old or above and indigenous people

Exclusion Criteria:

* Disability, have had oral cancer, impaired facial appearance and impaired cognitive function were excluded.

Impaired cognitive function was screening by Short Portable Mental Status Questionnaire (SPMSQ).

Ages: 55 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Oral health-related quality of life | Change from baseline at 3-month and 6-month after intervention
  OHRQoL was measured using the Geriatric Oral Health Assessment Index (GOHAI) , which was translated into Chinese for the participants (GOHAI-T). For example, "Are you satisfied or happy with the appearance of your teeth, gums or dentures?" Possible responses were range from 1 (always) to 5 (never). The total score ranged from 12 to 60 points. The higher the score, the better the quality of life. Cronbach's alpha was 0.75 for the scale.
Swallowing | Change from baseline at 2-week, 3-month and 6-month after intervention
  The Repetitive Saliva-Swallowing Test (RSST) was used to evaluate swallowing. Participants were asked to swallow saliva as many times as possible in 30 seconds.
syllable /pa/, /ta/ and /ka/ | Change from baseline at 2-week, 3-month and 6-month after intervention
  For oral diadochokinesis (DDK), the participants were asked to repeat the /pa/, /ta/, and /ka/ syllables as quickly as possible, and the number of articulations was counted. Using a digital counter, we separately counted the number of articulations of the /pa/, /ta/, and /ka/ syllables within 10 seconds.
Masticatory performance | Change from baseline at 2-week, 3-month and 6-month after intervention
  Masticatory performance was evaluated using the color-changeable chewing gum (Xylitol, 3.0 g Lotte, Saitama, Japan). This chewing gum contains xylitol, citric acid, and red, yellow, and blue dyes that change color when subjected to masticatory forces from chewing. The red dye is pH sensitive and changes color under neutral or alkaline conditions. Citric acid maintains a low internal pH of the yellowish-green gum before chewing commences. The gum changes to red when chewed because the yellow and blue dyes seep into saliva, and citric acid elution produces the red color. Participants were asked to chew for 2 minutes. Two minutes later, the observer checked the color of the gum by using a color chart of five color gradations ranging from 1 (very poor) to 5 (very good).
Saliva flow rate | Change from baseline at 2-week, 3-month and 6-month after intervention
  Saliva flow rate was measured the saliva flow rate in one minute (ml/min). Participants were asked to chew the gauze for two minutes and spited out the gauze and saliva back into the test tube. After centrifuging the saliva of the gauze, pour the saliva into a measuring tube to measure the volume of the saliva.
Perceived dysphagia | Change from baseline at 2-week, 3-month and 6-month after intervention
  Perceived dysphagia, which was defined as a subjective perception of problems swallowing, was measured using the swallowing screening scale developed by Ohkuma and has an internal consistency Cronbachα's alpha coefficient of 0.85. Examples of questions included "Do you ever have difficulty swallowing?" "Do you ever have difficulty as a result of cough up phlegm during or after a meal?" "Does it take you longer to eat a meal than it used to?" "Do you feel that it is becoming difficult to eat solid foods?" and "Do you ever have difficulty sleeping because of coughing during the night?" Possible responses were "obviously" (frequently), "slightly" (sometimes), or "no" (never). Respondents with at least one severe symptom were classified as having dysphagia.
Plaque control record (PCR) | Change from baseline at 2-week, 3-month and 6-month after intervention
  Plaque control record (PCR) was measured the percentage of tooth surface with plaque. PCR range from 0 to 100%.
Plaque index (PI) | Change from baseline at 2-week, 3-month and 6-month after intervention
  Plaque index (PI) was measured the six indicator teeth 12, 16, 24, 32, 36, 44 and the score for each tooth is range from 0 to 3 (0 = no plaque, 1 = a film of plaque adhering to the free gingival margin and adjacent area of the tooth, 2 = moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye, 3 = abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin). Then summing the average of 6 indicators teeth.
Winkel tongue coating index (WTCI) | Change from baseline at 2-week, 3-month and 6-month after intervention
  Winkel tongue coating index (WTCI) was measured the accumulation of coating on the surface of the tongue. The tongue was divided into six areas (three posterior and three anterior), and the coating was scored as 0 = no coating, 1 = light coating, or 2 = severe coating; scores ranged from 0 to 12 points.
Regular dental visit | Change from baseline at 2-week, 3-month and 6-month after intervention
  The question of dental visit, "Do you see a dentist every six months?" Possible responses were "Yes", "No".
Brushing ≥2 times/day | Change from baseline at 2-week, 3-month and 6-month after intervention
  The question of tooth-brushing, "How many times do you brush your teeth a day?" Possible responses were "None", "One time", "Two times" and "More than 3 times".
Use of interdental brushes | Change from baseline at 2-week, 3-month and 6-month after intervention
  The question of interdental brush, "Do you use an interdental brush every day?" Possible responses were "Yes", "No" and "Never heard".
Use of dental floss | Change from baseline at 2-week, 3-month and 6-month after intervention
  The question of flossing, "Do you use dental floss every day?" Possible responses were "Yes", "No" and "Never heard".

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Ling Huang, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT05046210/Prot_SAP_ICF_000.pdf